CLINICAL TRIAL: NCT06250205
Title: A Study to Evaluate the Effect of Daily Doses of Obicetrapib Tablets on the Pharmacokinetics of Drospirenone and Ethinyl Estradiol in Healthy Adult Female Subjects
Brief Title: Evaluate the Pharmacokinetics of a Combined Oral Contraceptive (COC) With and Without Obicetrapib
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NewAmsterdam Pharma (Industry)
Collaborators: Novum (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TA-8995-13
Record Dates: First submitted 2024-02-01; First posted 2024-02-08 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Healthy Volunteers
Keywords: DDI, drug-drug interaction, combined oral contraceptive
MeSH Terms: interventions — Tablets; drospirenone; Ethinyl Estradiol

STUDY DESIGN:
Intervention Model Description: Open-label, multiple-dose, fixed sequence, drug-drug interaction study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Treatment B+C: Obicetrapib + Drospirenone/Ethinyl Estradiol (COC) (Experimental): Obicetrapib 10 mg tablets and Drospirenone (3mg)/Ethinyl Estradiol (0.02mg) tablet
  Interventions: Drug: Obicetrapib; Drug: Obicetrapib + Drospirenone / Ethinyl Estradiol (COC)
- Treatment B: Obicetrapib (Experimental): Obicetrapib 10 mg tablets (daily)
  Interventions: Drug: Obicetrapib
- Treatment C: Drospirenone/Ethinyl Estradiol tablets (COC) (Experimental): Drospirenone (3mg)/Ethinyl Estradiol tablets (0.02mg) tablet
  Interventions: Drug: Drospirenone / Ethinyl Estradiol (COC)

INTERVENTIONS:
Drug: Obicetrapib — oral administration
  Other Names: 10 mg tablet
  Arms: Treatment B+C: Obicetrapib + Drospirenone/Ethinyl Estradiol (COC); Treatment B: Obicetrapib
Drug: Obicetrapib + Drospirenone / Ethinyl Estradiol (COC) — oral administration
  Other Names: tablets
  Arms: Treatment B+C: Obicetrapib + Drospirenone/Ethinyl Estradiol (COC)
Drug: Drospirenone / Ethinyl Estradiol (COC) — oral administration
  Other Names: tablets
  Arms: Treatment C: Drospirenone/Ethinyl Estradiol tablets (COC)

SUMMARY:
A study to evaluate the impact of Obicetrapib on the PK levels of Drospirenone and Ethinyl Estradiol (COC) in 30 adult female, healthy volunteers.

DETAILED DESCRIPTION:
This is an interventional, drug-drug interaction study to evaluate the effect of daily doses of Obicetrapib tablets on the pharmacokinetics of a combined oral contraceptive (COC), Drospirenone and Ethinyl Estradiol.

ELIGIBILITY:
Inclusion Criteria:

* Non-pregnant, non-lactating, non-tobacco-, non-nicotine-using female, 18-35 years of age, inclusive, who is a candidate for hormonal contraception (as determined by the Investigator).
* Subject has a BMI of 18.5-29.9 kg/m², inclusive. BMI will be calculated using Novum Pharmaceutical Research Services Standard Operating Procedures.
* If the subject is currently using a hormonal method of contraception, the subject is willing and agrees to stop using her hormonal contraceptive throughout the duration of the study and is prepared to abstain from sexual intercourse or use a reliable non-hormonal method of contraception, as outlined below

Exclusion Criteria:

* Male
* Have given birth or been pregnant within 3 months before initial dosing, or is currently pregnant, lactating or likely to become pregnant during the study.
* History of Hypertension, or seated blood pressure for a minimum of 5 minutes >140mmHg systolic, or > 80 mmHg, diastolic at screening

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2024-02-05 (Actual); Primary Completion 2024-04-25 (Actual); Study Completion 2024-04-26 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of COC | Upon completion of Treatment C (Day -6) and Treatments B+C (Day 12)
  Plasma Cmax concentration of COC with and without Obicetrapib
Area under the plasma concentration-time (AUC0-τ) curve for COC with and without coadministration with Obicetrapib | Upon completion of Treatment C (Day -6) and Treatments B+C (Day 12)
  Plasma AUC0-τ for COC with and without coadministration of Obicetrapib

CONTACTS AND LOCATIONS:
Overall Officials: Kent A Swaine, Principal Investigator — Novum Pharmaceutical Research Services, Inc.
Locations (1):
- NOVUM, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: No